CLINICAL TRIAL: NCT05547945
Title: The Effects of Health Promotion Program for the Caregivers of Attention Deficit/Hyperactivity Disorders Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Chang, Hsiu-Ju, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ADHD20180516
Record Dates: First submitted 2022-09-07; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: ADHD; Caregiver Stress Syndrome
Keywords: ADHD; Caregiver; Health Promotion Program
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Sixty caregivers were randomized to the health promotion group intervention (n=30) and the control groups (n=30). The control group received usual care.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This study used a randomized control trial design to perform simple sampling with using computer random sampling. Due to research recruitment, treatment intervention, and follow-up data tracking are different researchers, a single blind could reduce interference. The randomization procedure of this study was handled by the trained researcher. The researchers were responsible for different research interventions and data collection. The randomization of the password was not released during the study intervention to ensure the purpose of the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health promotion program (Other): The health promotion program included knowledge guidance on ADHD disease, physical activity, diet nutrition, parental training/stress adjustment, related social welfare resources, mindfulness relaxation, and yoga.
  Interventions: Behavioral: Health Promotion Program; Behavioral: Control group
- Control group (No Intervention): The control received as usual care.

INTERVENTIONS:
Behavioral: Health Promotion Program — The health promotion program included knowledge guidance on ADHD disease, physical activity, diet nutrition, parental training/stress adjustment, related social welfare resources, mindfulness relaxation, and yoga.
  Other Names: Experimental group
  Arms: health promotion program
Behavioral: Control group — The control group received as usual care.
  Other Names: Usual care
  Arms: health promotion program

SUMMARY:
Objective: To explore the effect of health promotion programs on parental stress, quality of life, and health-promoting lifestyles for primary caregivers who had children with ADHD. Children's ADHD symptoms were also examined.

Methods: A randomized control trial was conducted between July 2017 and April 2018. Primary caregivers aged 20 to 65 years who had ADHD children aged 7 to 12 years were recruited from a psychiatric outpatient department. Sixty caregivers were randomized to the health promotion group intervention (n=30) and the control groups (n=30). The control group received usual care. Study instruments included the Swanson, Nolan, Pelham, Version IV (SNAP-IV), Parenting Stress Scale (Short form), Taiwan's Concise World Health Organization Quality of Life Questionnaire (WHOQOL-BREF), and Health-Promotion Lifestyle Profile.

Both groups were evaluated before and immediately after the intervention at 1, 3, and 6 months. GEE was applied for statistical analysis.

Results: 60 participants were randomized to the health promotion intervention (n=30) or the control group (n=30). To explore the effect of health promotion programs on parental stress, quality of life, and health-promoting lifestyles for primary caregivers who are caring for children with ADHD.

Conclusion: We hope that the Health promotion program could demonstrate the effect in reducing parental stress, improving the quality of life, promoting healthy lifestyles for primary caregivers, and reducing the symptoms of children with ADHD. Proper intervention programs should be incorporated in clinical practice settings in order to facilitate mental health well-being for caregivers of ADHD children.

DETAILED DESCRIPTION:
Objective: To explore the effect of health promotion programs on parental stress, quality of life, and health-promoting lifestyles for primary caregivers who had children with ADHD. Children's ADHD symptoms were also examined.

Methods: A randomized control trial was conducted between July 2017 and April 2018. Primary caregivers aged 20 to 65 years who had ADHD children aged 7 to 12 years were recruited from a psychiatric outpatient department. Sixty caregivers were randomized to the health promotion group intervention (n=30) and the control groups (n=30). The control group received usual care. Study instruments included the Swanson, Nolan, Pelham, Version IV (SNAP-IV), Parenting Stress Scale (Short form), Taiwan's Concise World Health Organization Quality of Life Questionnaire (WHOQOL-BREF), and Health-Promotion Lifestyle Profile.

Both groups were evaluated before and immediately after the intervention at 1, 3, and 6 months. GEE was applied for statistical analysis.

Results: 60 participants were randomized to the health promotion intervention (n=30) or the control group (n=30). To explore the effect of health promotion programs on parental stress, quality of life, and health-promoting lifestyles for primary caregivers who are caring for children with ADHD.

Conclusion: We hope that the Health promotion program could demonstrate the effect in reducing parental stress, improving the quality of life, promoting healthy lifestyles for primary caregivers, and reducing the symptoms of children with ADHD. Proper intervention programs should be incorporated in clinical practice settings in order to facilitate mental health well-being for caregivers of ADHD children.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-65 years
* Being primary caregivers of children diagnosed with ADHD confirmed using DSM-IV aged 7-12 years
* Living together with the children and spending most of the time caring for children with ADHD among caregivers
* Being able to communicate by reading, listening and writing Chinese.

Exclusion Criteria:

* The primary caregivers who came to the out-patient department first time due to an undetermined diagnosis of ADHD
* Presence of the intellectual disability

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-19 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The Parenting Stress Scale (Short form) | 5 minutes
  Our study used a modified version of the parenting stress scale (Liu, 2015) which had 24 questions. The modified version of Abdin's short-term version of the parental stress scale is divided into three factors, including of parental distress, parent-child dysfunctional interaction, and difficult child.
The Taiwan's Concise World Health Organization Quality of Life Questionnaire (WHOQOL-BREF) | 5 minutes
  It had 28 questions, which are similar and well psychometrically measured to the global version of the questionnaire.
Health-Promotion Lifestyle Profile | 5minutes
  It has a total of 40 questions including of self-actualization, health-responsibility, exercise, nutrition, interpersonal support, stress management.

SECONDARY OUTCOMES:
ADHD symptoms | 5 minutes
  The Swanson, Nolan and Pelham, Version IV, SNAP-IV (Liu et al., 2006) The common version is a total of 26 questions for the SNAP-IV MTA, aged 6-13year-old children, including inattention subscales (1-9 questions), hyperactivity/impulse subscales (10-18 questions), and opposite subscales (19-26 questions).

CONTACTS AND LOCATIONS:
Locations (1):
- Wan Fang Hospital, Taipei Medical University, Taipei, Wenshan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Charach A, Carson P, Fox S, Ali MU, Beckett J, Lim CG. Interventions for preschool children at high risk for ADHD: a comparative effectiveness review. Pediatrics. 2013 May;131(5):e1584-604. doi: 10.1542/peds.2012-0974. Epub 2013 Apr 1. PMID 23545375